CLINICAL TRIAL: NCT00193232
Title: A Phase II Trial of Weekly Docetaxel and Bortezomib (Velcade; PS-341) in the Treatment of Patients With Advanced Hormone-Refractory Prostate Cancer
Brief Title: Weekly Docetaxel and Bortezomib in the Treatment of Advanced Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Aventis Pharmaceuticals (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GU 18; IIT16160
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Bortezomib

INTERVENTIONS:
Drug: Docetaxel
Drug: Bortezomib

SUMMARY:
Evaluation of the effectiveness of weekly docetaxel/bortezomib as first-line chemotherapy for patients with advanced hormone-refractory prostate cancer.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be receive:

* Docetaxel + Bortezomib

Patients with objective responses or stable disease will continue treatment for eight courses or until disease progression is documented.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer, and objective evidence of metastatic disease
* Progression while receiving androgen ablation therapy
* No previous chemotherapy
* Measurable or evaluable disease in conjunction with elevated serum PSA levels
* ECOG performance status 0, 1, or 2
* Adequate bone marrow, liver and kidney function
* Voluntarily provide written informed consent

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Moderate or severe peripheral neuropathy
* Age < 18 years
* Other serious medical conditions that may interfere with protocol therapy
* Other active malignancies
* history of treatment for other invasive cancers within 3 years

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-05; Primary Completion 2005-10 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
objective response rate

SECONDARY OUTCOMES:
progression-free survival
overall survival

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Hainsworth JD, Meluch AA, Spigel DR, Barton J Jr, Simons L, Meng C, Gould B, Greco FA. Weekly docetaxel and bortezomib as first-line treatment for patients with hormone-refractory prostate cancer: a Minnie Pearl Cancer Research Network phase II trial. Clin Genitourin Cancer. 2007 Mar;5(4):278-83. doi: 10.3816/CGC.2007.n.004. PMID 17553208
- See also: Published article in Clinical Genitourinary Cancer — http://cigjournals.metapress.com/content/628584521732211v/?p=9226ef7cd8ae499bae10afa2132095c7&pi=4